CLINICAL TRIAL: NCT03517982
Title: MyOra® (Mycophenolate Mofetil) Post-Authorization Safety Study for Prophylaxis in de Novo Renal Transplant Patients
Brief Title: Generic Mycophenolate Mofetil Safety Study for Prophylaxis in de Novo Renal Transplant Patients in Jordan
Acronym: MyOra-PASS
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MYR-JOR-2013-04
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Acute Transplant Rejection in Patients Receiving Allogeneic Renal Transplant
Keywords: MyOra; Mycophenolate Mofetil; End stage renal disease; De novo Renal transplant; Post authorization safety study; Immunosuppressant; Cohort study
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Film Coated Tablet, each tablet contains 500mg Mycophenolate Mofetil
  Other Names: MyOra®

SUMMARY:
The purpose of this observational study was to assess the safety and efficacy of generic mycophenolate mofetil in de novo renal transplant patients in Jordan where no visits or intervention(s) additional to the daily practice were performed.

DETAILED DESCRIPTION:
A single center, observational, open-label, longitudinal, prospective study combined with retrospective data collection for 12 de novo renal transplant patients. Ten patients were prospectively followed for 12 months after receiving MyOra® (mycophenolate mofetil) and two patients were previously on MyOra® (mycophenolate mofetil), thus their data was retrospectively collected from their hospital records and all relevant workup tests results. Outcomes include occurrence of AEs and proportion of patients with normal graft function.

ELIGIBILITY:
Inclusion Criteria:

* Patient received de novo renal transplant
* Patient treated with MyOra® according to the attending physician's judgment (either post-transplant or induction)
* Patient provided written informed consent

Exclusion Criteria:

* Hypersensitivity to mycophenolate mofetil, mycophenolic acid (MPA) or any of the constituents of MyOra®

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients were enrolled from a single public hospital in Jordan
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of adverse events (AEs) to the Study medication | 12 months
  Rate of AEs, SAEs and laboratory tests abnormalities will be calculated

SECONDARY OUTCOMES:
Proportion of patients with normal graft function | 12 months
  Graft status was estimated through the evaluation of kidney function in all patients enrolled in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Hamza Hospital, Amman, Jordan